CLINICAL TRIAL: NCT05194137
Title: Biofeedback Versus Vaginal Palpation to Teach a Voluntary Pelvic Floor Muscle Contraction to Women Incapable of Performing it? A Non-inferiority Randomized Controled Trial
Brief Title: Biofeedback Versus Vaginal Palpation to Teach a Voluntary Pelvic Floor Muscle Contraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, ANA CAROLINA NOCITI LOPES FERNANDES, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32215720.0.0000.5440
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: The randomization of the participants will be done using a computer-generated list of numbers (www.randomization.com). This list will be put in a sealed envelope and participants allocation will be concealed.
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for assessment and inclusion of participants in the study will be blinded to which group participants will be allocated to. The research assistant who is responsible for generate the list of randomized numbers and seal the envelope as well as the research assistant responsible to perform patients' allocation will not be involved in the recruitment, assessment of participants or interventions.
  Blinding of participants, and treatment providers: not possible Blinding of outcome measurement: Primary outcome - blinded assessment by a physiotherapist not involved in delivery of therapy or with knowledge of group allocation. All other outcomes - not blinded because they are patient-reported.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a proprioception protocol associated with vaginal palpation and feedback (CG) (Active Comparator): The participants of CG will be placed in the supine position with flexion of the hip and knee and feet supported on the stretcher. Vaginal palpation will be used as a proprioceptive resource to facilitate PFM voluntary contraction. The physiotherapist responsible for conducting the treatment, wearing gloves, will perform a one or two-finger vaginal palpation, depending on participant's vaginal canal.
  Positive reinforcements will be verbalized after each PFM contraction. The training protocol will be tailored, and the evolution will be the same for CG and BPFMT.
  Interventions: Other: a proprioception protocol associated with vaginal palpation and feedback
- a proprioception protocol associated with biofeedback (BG) (Experimental): The participants of BG will receive the same protocol of CG but associated with biofeedback with an electromyographic sensor through the Miotol equipment (Miotec, Brazil). The participants of the BG will also be positioned in the same position described to CG. The electromyographic sensor will be covered with neutral gel and inserted into the participant's vaginal canal. Participants will see the visual response of the contraction on the computer screen. The software has five different interfaces for visualize PFM contraction and each participant will be able to choose the one that she prefers at each session. The training protocol will be tailored, and the evolution will be the same for CG and BG. During the first session, it will be explained what is biofeedback and what means everything that appears on the software interface.
  Interventions: Other: a proprioception protocol associated with biofeedback

INTERVENTIONS:
Other: a proprioception protocol associated with vaginal palpation and feedback — A total of 13 previously established examples of voice commands can be used by the physiotherapists to help women understand how to perform a PFM contraction.
  Arms: a proprioception protocol associated with vaginal palpation and feedback (CG)
Other: a proprioception protocol associated with biofeedback — The software has five different interfaces for visualize PFM contraction: sign itself and signal transformed into the movement of a balloon; an airplane; a fairy; or a bird. Positive reinforcements will be verbalized after each PFM contraction using one of 4 previously established examples of voice commands.
  Arms: a proprioception protocol associated with biofeedback (BG)

SUMMARY:
Pelvic floor muscle training (PFMT) is the first line treatment of urinary incontinence (UI), anal incontinence (AI) and mild/moderate pelvic organ prolapse (POP) in women. However, 25 to 40% of women with pelvic floor dysfunction symptoms are unable to voluntarily contract their pelvic floor muscle (PFM) and PFM proprioception of this population is specially reduced. Literature is scarce about methods to facilitate a voluntary PFM contraction and improve PFM proprioception therefore, a specific protocol structured to teach PFM contraction is needed. The use of biofeedback could facilitate women´s capacity to voluntary contract their PFM.

DETAILED DESCRIPTION:
Randomised, parallel (two arm), trial comparing biofeedback (experimental arm) versus vaginal palpation (active control, i.e. usual practice) to achieve a correct voluntary pelvic floor muscle contraction in women who cannot perform a correct contraction (i.e. grade 0, 1 or 2 on the Modified Oxford Scale). The trial hypothesis is that there is no difference between the two trial arms in the proportion of women achieving a correct voluntary contract (grade 3 or better).

The training protocol will be the same for both groups and will vary according to PFM function assessed at 0, 3, 6 and 9-week timepoint. The resting time after each contraction will be the double of the contraction duration, therefore if it is performed a 3-second contraction, it will be a 6-second rest. The first session will aim to improve some skills as understanding, searching, and finding PFM, the educational component of this session was structured considering Health Belief Model and will be conducted with the following information: 1) General information (female genital anatomy, female intern organs, pelvic floor muscle anatomy, pelvic floor muscle function), 2) specific information about urinary incontinence (definition of urinary incontinence, predictors of risk for urinary incontinence, impact on quality of life), 3) the relation between PFM and urinary incontinence, 4) pelvic floor muscle training as first line treatment for urinary incontinence, 5) how to include PFM proprioception protocol into daily life. It will be used as educational materials images and draws of the region and an educational booklet will be delivered to them. It will be shown to then a video of a PFM contraction emphasizing how the correct PFM contraction is supposed to be. The other sessions will focus will vary according to PFM function accessed at each timepoint:

* Participants classified with MOS 0 or 1: PFM protocol will aim on learning a PFM contraction and improve PFM perception
* Participants classified with MOS = 2: PFM protocol will aim on teaching how to control PFM contraction
* Participants classified with MOS ≥ 3: PFM protocol will aim on improving PFM strength

The resting time after each set will be 3 minutes and the protocol will evolve as following:

* WEEK 1: In clinics: 30 minutes: educational component as previous discussed. 30 minutes: The studied protocol will be explained as well as the need to fulfill a diary with their home training routine that should be delivered to the evaluator at the 12-week assessment. At each session, the physiotherapist will oversee the diary, take notes about the frequency of training, and orientate if necessary. To promote a first contact with their PFM, it will be performed 1 set of PFM contraction associated with vaginal palpation or biofeedback of 6 fast contraction according to the randomized group. The resting time after each contraction will be five seconds. Possible doubts will be clarified. At home: All participants will be oriented to perform 3 sets of 6 fast contraction daily during the following week in the supine position. The resting time after each contraction will be five seconds and after each set will be 2 minutes.
* WEEK 2-3: In clinics: Training diary will be overseen, and possible doubts will be clarified. Training protocol will be different according to PFM function assessed on week 0. MOS 0: 3 sets of 6 fast contraction. The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 6 fast contraction and 3 sets of 6 contractions sustained for 3 seconds. The resting time after each contraction will be five seconds and 2 minutes after each set. At home: Training protocol will be different according to PFM function assessed on week 0. MOS 0: 3 sets of 6 fast contraction in supine position. The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 6 fast contraction and 3 sets of 6 contractions sustained for 3 seconds in supine. The resting time after each contraction will be five seconds and 2 minutes after each set.
* WEEK 4-6: In clinics: Training diary will be overseen, and possible doubts will be clarified. Training protocol will be different according to PFM function assessed on week 3. MOS 0: 3 sets of 10 fast contraction. The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 10 fast contraction and 3 sets of 6 contractions sustained for 4 seconds. The resting time after each contraction will be six seconds and 2 minutes after each set. MOS ≥ 2: 3 sets of 10 fast contraction and 3 sets of 10 contractions sustained for 6 seconds. The resting time after each contraction will be ten seconds and 3 minutes after each set. At home: Training protocol will be different according to PFM function assessed on week 3. MOS 0: 3 sets of 10 fast contraction, each set on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 10 fast contraction and 3 sets of 6 contractions sustained for 4 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be six seconds and 2 minutes after each set. MOS ≥ 2: 3 sets of 10 fast contraction and 3 sets of 10 contractions sustained for 6 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be ten seconds and 3 minutes after each set.
* WEEK 7-9: In clinics: Training diary will be overseen, and possible doubts will be clarified. Training protocol will be different according to PFM function assessed on week 6. MOS 0: 3 sets of 10 fast contraction and 3 sets of 5 contraction sustained for 3 seconds. The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 10 fast contraction and 3 sets of 6 contractions sustained for 4 seconds. The resting time after each contraction will be six seconds and 2 minutes after each set. MOS ≥ 2: 3 sets of 10 fast contraction and 3 sets of 10 contractions sustained for 6 seconds. The resting time after each contraction will be ten seconds and 3 minutes after each set. At home: Training protocol will be different according to PFM function assessed on week 6. MOS 0: 3 sets of 10 fast contraction and 3 sets of 5 contraction sustained for 3 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 10 fast contraction and 3 sets of 6 contractions sustained for 4 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be six seconds and 2 minutes after each set. MOS ≥ 2: 3 sets of 10 fast contraction and 3 sets of 10 contractions sustained for 6 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be ten seconds and 3 minutes after each set.
* WEEK 10-12: In clinics: Training diary will be overseen, and possible doubts will be clarified. Training protocol will be different according to PFM function assessed on week 9. MOS 0: 3 sets of 10 fast contraction and 3 sets of 5 contraction sustained for 3 seconds. The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 10 fast contraction and 3 sets of 6 contractions sustained for 4 seconds. The resting time after each contraction will be six seconds and 2 minutes after each set. MOS ≥ 2: 3 sets of 10 fast contraction and 3 sets of 10 contractions sustained for 6 seconds. The resting time after each contraction will be ten seconds and 3 minutes after each set. At home: Training protocol will be different according to PFM function assessed on week 6. MOS 0: 3 sets of 10 fast contraction and 3 sets of 5 contraction sustained for 3 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be five seconds and after each set will be 2 minutes. MOS 1: 3 sets of 10 fast contraction and 3 sets of 6 contractions sustained for 4 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be six seconds and 2 minutes after each set. MOS ≥ 2: 3 sets of 10 fast contraction and 3 sets of 10 contractions sustained for 6 seconds. Each set is supposed to be performed on a different position (i.e. supine, sitting and standing). The resting time after each contraction will be ten seconds and 3 minutes after each set.

The two groups will receive a booklet and guidance to perform the training protocol at home on alternate days and a diary to register their adherence to the program. The guided protocol will be the same used during the supervised training on that specific week. Women will be oriented to choose the position to practice unsupervised sessions (i.e. supine,lateral, sitting and/or standing).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or over;
* Women referred to the physiotherapeutic treatment of the Lucy Montoro Rehabilitation Center (Ribeirão Preto Medical School) or the Women's Health Reference Center (MATER) for any pelvic floor dysfunction;
* Women unable to perform a PFM contraction (i.e. PFM function classified as 0 or 1 according to the modified oxford scale);
* Women with urinary incontinence (i.e ICIQ-UI-SF score ≥ 3)
* Agree to participate in the research by signing the informed consent form

It will not be included in this study:

* Women whose pelvic floor dysfunction has an associated neuropathy;
* Women with vaginal or urological symptoms of possible infections;
* Women with pelvic organs prolapse that makes it impossible to evaluate or conduct treatment (stage > 2 according to Baden-Walker Scale);
* Pregnant women;
* Women with cognitive impairment.

Exclusion Criteria:

* Women who become pregnant while conducting the study
* Women with intolerance or pain that prevents the conduct of research protocols.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
change in ability to perform a voluntary PFM contraction | At baseline, 3, 6, 9 and 12 weeks
  be to gain the ability to perform a voluntary PFM contraction assessed by vaginal palpation and classified by the modified oxford scale (MOS). Women able to perform PFM contraction with both occlusion of the vaginal opening and inward movement will be considered able to perform a voluntary PFM contraction, this is the description of MOS grade 3.

SECONDARY OUTCOMES:
Urinary incontinence (UI) | baseline and 12 weeks
  The presence of UI, its severity and impact on quality of life will be assessed by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-UI-SF)
self-perception of pelvic floor muscle (PFM) contraction | At baseline, 3, 6, 9 and 12 weeks
  Self-perception of PFM contraction will be a self-reported measure classified according to Modified oxford scale (MOS). MOS is a categorical variable with 6 possible answers ranging from 0 to 5.
adherence to treatment | weekly up to 12 weeks
  Adherence to supervised and unsupervised treatment will be assessed with physiotherapist registration of sessions and participants' exercise diary respectively. This is a descriptive variable that will range from 0 to 12 sessions (supervised treatment) and from 0 - 36 days (unsupervised treatment).
adverse effects | 12 weeks
  Adverse effects will be assessed using the following question "Did you experienced any discomfort or warm during supervised treatment?" at the lest assessment timepoint.
satisfaction with treatment | 12 weeks
  Satisfaction with treatment will be assessed using a numerical scale (0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05194137/Prot_001.pdf